CLINICAL TRIAL: NCT00724958
Title: Real Life Dosing Regimen of Remicade in Austria in Crohn's Disease - Program Extension
Brief Title: Program Extension of Real Life Dosing of Remicade in Austria for Crohn's Disease (Study P04052)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: P04052
Record Dates: First submitted 2008-07-25; First posted 2008-07-30 (Estimated); Results first posted 2011-10-26 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Remicade: Subjects with active luminal and/or fistulizing CD in the hospital or non-hospital setting.
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: Infliximab — Not specified in the protocol.
  Other Names: Remicade; SCH 215596

SUMMARY:
The current observational program was determined to collect data on the real life dosing regimen of Remicade in patients with Crohn's disease (CD) in the hospital and non-hospital setting.

DETAILED DESCRIPTION:
This study population was chosen from a non-probability sample

ELIGIBILITY:
Inclusion Criteria:

* Subjects with active luminal and/or fistulizing CD.

Exclusion Criteria:

* Per summary of product characteristics.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with active luminal and/or fistulizing CD who are treated with Remicade in the hospital and non-hospital setting.
Sampling Method: Non-Probability Sample
Enrollment: 348 (Actual)
Dates: Start 2004-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Remicade: Subjects with active luminal and/or fistulizing Crohn's Disease in the hospital or non-hospital setting.
Period: Overall Study
Arm/Group | Remicade
Started | 348
Completed | 166
Not Completed | 182
Not completed — Adverse Event | 28
Not completed — Loss of Response | 40
Not completed — No Response | 18
Not completed — Remission | 7
Not completed — Other Reason | 76
Not completed — No documentation for end of therapy | 13

BASELINE CHARACTERISTICS:
Groups:
- Remicade: Subjects with active luminal and/or fistulizing Crohn's Disease in the hospital or non-hospital setting who received at least one infliximab infusion.
Arm/Group | Remicade
Number analyzed (Participants) | 343
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.68 (12.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178
  Male | 165
Region of Enrollment [Number; unit: participants]
  Austria | 343

OUTCOME MEASURES:

1. Primary Outcome: Mean Interval Between Infliximab Infusions Within the Observation Period (Maintenance Therapy)
Description: Participants received infliximab infusions with or without induction therapy. The induction therapy consisted of three infliximab infusions at Weeks 0, 2 and 6. Maintenance therapy consisted of an additional 6 infusions (maximum) as prescribed by the treating physician (dose and infusion interval).
Time Frame: up to 2 years
Population: n = number of infliximab-naive participants
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Remicade
Number analyzed (Participants) | 298
Days
  Interval between infusion 1 & 2, n=298 | 16.89 (11.35)
  Interval between infusion 2 & 3, n=275 | 34.74 (17.14)
  Interval between infusion 3 & 4, n=250 | 63.22 (26.07)
  Interval between infusion 4 & 5, n=227 | 62.86 (26.40)
  Interval between infusion 5 & 6, n=210 | 61.30 (18.03)
  Interval between infusion 6 & 7, n=186 | 60.95 (20.16)
  Interval between infusion 7 & 8, n=162 | 59.24 (16.81)
  Interval between infusion 8 & 9, n=148 | 60.22 (16.55)

2. Primary Outcome: Median Interval Between Infliximab Infusions Within the Observation Period (Maintenance Therapy)
Description: as for outcome 1
Time Frame: up to 2 years
Population: n = number of infliximab-naive participants
Measure: Median (Full Range); unit: Days
Arm/Group | Remicade
Number analyzed (Participants) | 298
Days
  Interval between infusion 1 & 2, n=298 | 14.00 [5 to 129]
  Interval between infusion 2 & 3, n=275 | 28.00 [11 to 182]
  Interval between infusion 3 & 4, n=250 | 56.00 [18 to 266]
  Interval between infusion 4 & 5, n=227 | 57.00 [14 to 273]
  Interval between infusion 5 & 6, n=210 | 57.00 [23 to 184]
  Interval between infusion 6 & 7, n=186 | 56.00 [24 to 214]
  Interval between infusion 7 & 8, n=162 | 56.00 [15 to 161]
  Interval between infusion 8 & 9, n=148 | 56.00 [11 to 140]

3. Secondary Outcome: Assessment of the Disease Activity Before Treatment and During Therapy With Remicade Via Harvey Bradshaw Index (HBI) in an Extended Patient Group of 200 Patients.
Description: HBI consists of only clinical parameters (general well-being, abdominal pain, number of liquid stools per day, abdominal mass, and complications). HBI is a score on a scale; <5 (remission), 5-7 (mild disease), 8-16 (moderate disease), >16 (severe disease).
Time Frame: 5 years
Population: 207 participants had disease activity analyzed using Harvey-Bradshaw Index (HBI)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Remicade
Number analyzed (Participants) | 207
Score on a scale
  Infusion 1, n=44 | 8.25 (5.60)
  Infusion 2, n=28 | 3.46 (3.69)
  Infusion 3, n=19 | 2.21 (2.04)
  Infusion 4, n=20 | 2.40 (2.85)
  Infusion 5, n=23 | 2.70 (3.36)
  Infusion 6, n=24 | 3.38 (4.19)
  Infusion 7, n=17 | 2.06 (2.05)
  Infusion 8, n=17 | 2.29 (2.62)
  Infusion 9, n=15 | 2.67 (2.89)

4. Primary Outcome: Average Dose of Infliximab Per Participant Within the Observation Period
Description: as for outcome 1
Time Frame: up to 2 years
Population: n = number of infliximab-naive participants
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Remicade
Number analyzed (Participants) | 315
mg/kg
  Infusion 1, n=315 | 5.09 (0.66)
  Infusion 2, n=300 | 5.04 (0.67)
  Infusion 3, n=276 | 5.06 (0.62)
  Infusion 4, n=253 | 5.11 (0.76)
  Infusion 5, n=227 | 5.20 (1.02)
  Infusion 6, n=210 | 5.17 (0.95)
  Infusion 7, n=186 | 5.19 (0.92)
  Infusion 8, n=163 | 5.22 (1.03)
  Infusion 9, n=148 | 5.25 (0.97)

5. Primary Outcome: Median Dose of Infliximab Per Participant Within the Observation Period
Description: as for outcome 1
Time Frame: up to 2 years
Population: n = number of infliximab-naive participants
Measure: Median (Full Range); unit: mg/kg
Arm/Group | Remicade
Number analyzed (Participants) | 315
mg/kg
  Infusion 1, n=315 | 5.09 [2.56 to 8.62]
  Infusion 2, n=300 | 5.00 [2.31 to 8.77]
  Infusion 3, n=276 | 5.00 [3.19 to 8.77]
  Infusion 4, n=253 | 5.00 [3.66 to 11.43]
  Infusion 5, n=227 | 5.00 [3.64 to 11.43]
  Infusion 6, n=210 | 5.00 [3.41 to 11.36]
  Infusion 7, n=186 | 5.08 [3.41 to 11.43]
  Infusion 8, n=163 | 5.10 [3.41 to 11.11]
  Infusion 9, n=148 | 5.12 [3.37 to 9.84]

6. Primary Outcome: Total Dose of Infliximab Per Participant Within the Observation Period
Description: as for outcome 1
Time Frame: up to 2 years
Population: 315 of infliximab-naive participants were treated in the active phase of the study. Of these, 191 participants received induction therapy (Weeks 0, 2, and 6); 27 received only induction therapy, 132 received induction therapy and subsequent maintenance therapy, and 32 received induction therapy and subsequent episodic therapy.
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Remicade
Number analyzed (Participants) | 315
mg/kg | 2290.32 (1096.04)

ADVERSE EVENTS:
Arm/Group | Remicade
Serious Adverse Events (participants affected / at risk) | 43/343
Other Adverse Events (participants affected / at risk) | 0/343
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remicade (N=343)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1)
Colonic Stenosis (Gastrointestinal disorders) | 1 (1)
Crohn's Disease (Gastrointestinal disorders) | 1 (1)
Ileal Stenosis (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Intestinal Perforation (Gastrointestinal disorders) | 1 (1)
Small Intestinal Stenosis (Gastrointestinal disorders) | 2 (2)
Subileus (Gastrointestinal disorders) | 2 (4)
Anaphylactic Reaction (Immune system disorders) | 2 (2)
Cytokine Release Syndrome (Immune system disorders) | 1 (1)
Drug Hypersensitivity (Immune system disorders) | 2 (2)
Abscess (Infections and infestations) | 3 (3)
Anal Abscess (Infections and infestations) | 2 (2)
Herpes Virus Infection (Infections and infestations) | 1 (1)
Nasal Abscess (Infections and infestations) | 1 (1)
Perirectal Abscess (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Aspiration Bone Marrow (Investigations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
B-cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cluster Headache (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Simple Partial Seizures (Nervous system disorders) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Abscess Drainage (Surgical and medical procedures) | 4 (4)
Appendicectomy (Surgical and medical procedures) | 1 (1)
Colectomy (Surgical and medical procedures) | 1 (1)
Enterostomy (Surgical and medical procedures) | 1 (1)
Enterostomy Closure (Surgical and medical procedures) | 1 (1)
Hospitalization (Surgical and medical procedures) | 3 (3)
Intestinal Operation (Surgical and medical procedures) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No